CLINICAL TRIAL: NCT00600652
Title: Flow Cytometric Analysis of Glucocorticoid Receptor Using Monoclonal Antibody and Fluoresceinated Ligand Probes in Glucocorticoid-Resistant and -Sensitive Patients
Brief Title: FCM Analysis GR in Steroid-Treatment Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Changhai Hospital (Other)
Responsible Party: ChangQuan Ling, Department of integrative medicien,Changhai Hospital
Other Study IDs: 061210; 30730114
Record Dates: First submitted 2008-01-15; First posted 2008-01-25 (Estimated); Last update posted 2008-01-25 (Estimated); Status verified 2008-01

CONDITIONS: Healthy
Keywords: glucocorticoid-receptor; flow cytometry; glucocorticoid-resistant; prediction

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — introcellular and exocellular proteins in peripheral blood mononuclear cells of subjects
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: glucocorticoid-resistant patients
- 2: glucocorticoid-sensitive patients
- 3: normal controls

SUMMARY:
Monitoring the GR with a GR-MoAb and FITC-Dex probes by FCM would be useful and convenient in determination GR before the steroid treatment in clinical, especially in steroid resistant states, in order to design more efficient clinical treatment protocols.

DETAILED DESCRIPTION:
In order to assess the efficacy of this method, 100 patients with nephrotic syndrome and systemic lupus erythematosus receiving sufficient prednisolone thereafter and 50 age- and sex-matched normal controls will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of SLE and NS

Exclusion Criteria:

* Receiving hormone replacement therapy or had received hormone replacement therapy in three months before start of the study
* Received drugs or drinks containing alcohol within one month
* Having symptom such as infection
* Supersensitivity and endocrine disturbance.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: one hundred patients, including 50 SLE and 50 NS, who will receive GC therapy, were studied. Of them, fifty were GC-resistant patients (25 male and 25 female; 20 without treatment and 30 relapse) and fifty were GC-sensitive ones( 25 male and 25 female; 20 without treatment and 30 relapse ). Controls were 50 healthy volunteers (25 male and 25 female). All participants gave their informed consent, and this investigation was approved by Changhai hoapital ethics committee.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2006-12; Primary Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jing Li, professor, Principal Investigator — Changhai Hospital

REFERENCES:
- [Derived] Du J, Li M, Zhang D, Zhu X, Zhang W, Gu W, Feng Y, Zhai X, Ling C. Flow cytometry analysis of glucocorticoid receptor expression and binding in steroid-sensitive and steroid-resistant patients with systemic lupus erythematosus. Arthritis Res Ther. 2009;11(4):R108. doi: 10.1186/ar2763. Epub 2009 Jul 14. PMID 19594946